CLINICAL TRIAL: NCT04189094
Title: Chemoradiotherapy With or Without Sintilimab in Limited-stage Small Cell Lung Cancer: a Multicenter Prospective Randomized Phase II Trial
Brief Title: Chemoradiotherapy With or Without Sintilimab in Limited-stage SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Hospital of Guangdong Medical University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2019-164
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: radiotherapy; chemotherapy; immunotherapy; PD-1 inhibitor; lung cancer; small cell; limited-stage
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; Etoposide; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab + CRT arm (Experimental): Patients with limited-stage SCLC receive etoposide and cisplatin (carboplatin) plus Sintilimab induction therapy for 2 cycles and then receive thoracic radiotherapy (45 Gy/30 fractions) with concurrent EP/EC chemotherapy for 2cycles. Patients who achieve CR or PR then receive prophylactic cranial irradiation (PCI, 25 Gy/10 fractions). After PCI, Sintilimab maintenance therapy will be administered once every 3 week for 13 cycles.
  Interventions: Drug: Sintilimab; Drug: Etoposide; Drug: Cisplatin; Radiation: radiotherapy
- CRT arm (Active Comparator): Patients with limited-stage SCLC receive etoposide and cisplatin (carboplatin) for 2 cycles and then receive thoracic radiotherapy (45 Gy/30 fractions) with concurrent EP/EC chemotherapy for 2cycles. Patients who achieve CR or PR then receive prophylactic cranial irradiation (PCI, 25 Gy/10 fractions).
  Interventions: Drug: Etoposide; Drug: Cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Etoposide and cisplatin (carboplatin) plus Sintilimab induction therapy will be administered for 2 cycles and then thoracic radiotherapy (45 Gy/30 fractions) be administered with concurrent EP/EC chemotherapy for 2cycles. Patients who achieve CR or PR then receive prophylactic cranial irradiation (PCI, 25 Gy/10 fractions).Sintilimab maintenance therapy will be administered once every 3 week for 13 cycles.
  Arms: Sintilimab + CRT arm
Drug: Etoposide — Etoposide will be administered IV 100mg/m2 on days 1-3, 22-24, 43-45 and 64-66.
  Other Names: VP-16
Drug: Cisplatin — cisplatin will be administered IV 80mg/m2 on days 1, 22, 43 and 64.
  Other Names: DDP
Radiation: radiotherapy — Thoracic radiotherapy (45 Gy/30 fractions) and prophylactic cranial irradiation (25 Gy/10 fractions).

SUMMARY:
The study is a prospective, multi-center, open-label, randomized, and controlled phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed diagnosis of SCLC.
2. Radiologically (including brain CT/MRI, chest and abdomen contrasted CT and bone scintigraphy. PET/CT is recommended) confirmed limited-stage.
3. Patients should be ≥ 18 years old.
4. ECOG performance status of 0-1 (Karnofsky performance status ≥ 80).
5. With adequate cardiac, pulmonary, bone marrow, hepatic and renal function.
6. With weight loss no more than 10% within 6 months before diagnosis.
7. Informed consent must be signed.

Exclusion Criteria:

1. Histology confirmed the mixed NSCLC components;
2. Other primary malignant tumors appeared within 5 years before the first administration of the study drug, except for locally curable malignant tumors after radical treatment (such as basal or squamous cell skin cancer, superficial bladder cancer or prostate, cervical or breast carcinoma in situ, etc.);
3. Any disease or condition contraindicated by radiotherapy or chemotherapy;
4. Malignant pleural effusion and pericardial effusion;
5. Pregnant and lactating women;
6. History of idiopathic pulmonary fibrosis (IPF), including pneumonia and organic pneumonia;
7. Received live vaccination within 28 days before the first administration of the study drug;
8. 28 days prior to the first administration of the study drug, he participated in any other drug clinical trials or is undergoing other clinical trials.
9. Have received any antibody / drug (including PD-1, PDL1, CTLA4, tim3, Lag3, etc.) targeting T-cell co regulatory protein (immunocheckpoint).
10. The investigator believes that the subject's complications or other circumstances may affect the compliance with the protocol or may not be suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  PFS, defined as the time from the date of randomization to the first date of documented objective progression disease or of death from any cause.

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS, measured from the date of randomization to the date of death from any cause.
Overall response rates | 2 years
  ORR, tumor response will be measured by using the RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, MD. PhD., Principal Investigator — Cancer Hospital of the University of Chinese Academy of Science (Zhejiang Cancer Hospital)